CLINICAL TRIAL: NCT03611751
Title: A Multi-Center, Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Phase 3 Study With Randomized Withdrawal and Retreatment to Evaluate the Efficacy and Safety of BMS-986165 in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: An Investigational Study to Evaluate Experimental Medication BMS-986165 Compared to Placebo and a Currently Available Treatment in Participants With Moderate-to-Severe Plaque Psoriasis
Acronym: POETYK-PSO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-047; 2018-001925-24 (EudraCT Number)
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib; apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986165 (Experimental): BMS-986165 oral administration
  Interventions: Drug: BMS-986165
- Placebo (Placebo Comparator): Placebo oral administration
  Interventions: Other: Placebo
- Active comparator (Active Comparator): Active comparator oral administration
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Arms: BMS-986165
Other: Placebo — Specified dose on specified days
  Arms: Placebo
Drug: Apremilast — Specified dose on specified days
  Arms: Active comparator

SUMMARY:
The purpose of this study is to investigate the experimental medication BMS-986165 compared to placebo and a currently available treatment in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Plaque psoriasis for at least 6 months
* Moderate to severe disease
* Candidate for phototherapy or systemic therapy

Exclusion Criteria:

* Other forms of psoriasis
* History of recent infection
* Prior exposure to BMS-986165 or active comparator

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (205):
- United States (89):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - Alliance Dermatology and Mohs Center - Phoenix, Phoenix, Arizona
  - Clinical Research Consortium - Tempe, Tempe, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Associates in Research, Inc., Fresno, California
  - Marvel Clinical Research, Huntington Beach, California
  - Interspond - Long Beach Clinical Trials, Long Beach, California
  - Dermatology Research Associates - Los Angeles, Los Angeles, California
  - LA Universal Research Center, Los Angeles, California
  - Artemis Institute for Clinical Research - San Diego, San Diego, California
  - University of California San Diego Health Systems, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - San Luis Dermatology and Laser Clinic, San Luis Obispo, California
  - Artemis Institute for Clinical Research - San Marcos, San Marcos, California
  - West Coast Research, San Ramon, California
  - Clinical Science Institute, Santa Monica, California
  - Synexus - Santa Rosa, Santa Rosa, California
  - Care Access Research - Walnut Creek, Walnut Creek, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Skin Care Research, Boca Raton, Florida
  - ERN - Accel Research - Avail, DeLand, Florida
  - Interspond - Savin Medical Group, Miami Lakes, Florida
  - Synexus Clinical Research - Saint Petersburg, Pinellas Park, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Precision Clinical Research - Corporate Office, Sunrise, Florida
  - Precision Clinical Research - Corporate Office, Tamarac, Florida
  - Moore Clinical Research - South Tampa, Tampa, Florida
  - University of South Florida/USF Health, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Marietta Dermatology & The Skin Cancer Center, Marietta, Georgia
  - Advanced Clinical Research - Idaho, Meridian, Idaho
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dermatology Center of Northwest Indiana, Crown Point, Indiana
  - Synexus - Evansville South, Evansville, Indiana
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - Skin Sciences, Louisville, Kentucky
  - Advanced Medical Research, Lacombe, Louisiana
  - Shondra L. Smith, M.D., Lake Charles, Louisiana
  - DelRicht Research - New Orleans - Prytania Street, New Orleans, Louisiana
  - Ora, Andover, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham Dermatology Associates, Boston, Massachusetts
  - A. Alfred Taubman Health Care Center, Ann Arbor, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Washington University School of Medicine - West County Dermatology, Creve Coeur, Missouri
  - Healthcare Research Network - Hazelwood, Hazelwood, Missouri
  - Clinical Research Consortium - Las Vegas, Las Vegas, Nevada
  - ActivMed Practices and Research - Portsmouth, Portsmouth, New Hampshire
  - Windsor Dermatology, East Windsor, New Jersey
  - Sadick Research Group, New York, New York
  - DermResearch Center of New York, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - PMG Research of Cary, Cary, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Synexus - Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Wright State Research Institute, Fairborn, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology and Skin Surgery Center - Exton, Exton, Pennsylvania
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - Synexus, Greer, South Carolina
  - Coastal Carolina Research Center - Mount Pleasant, Mt. Pleasant, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Rivergate Dermatology - Main Office, Goodlettsville, Tennessee
  - Clinical Research Solutions - Jackson, Jackson, Tennessee
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - The Skin Wellness Center, Knoxville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - DermResearch, Austin, Texas
  - Bellaire Dermatology, Bellaire, Texas
  - Modern Research Associates, Dallas, Texas
  - Synexus - Dallas, Dallas, Texas
  - Progressive Clinical Research - San Antonio, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Interspond - Houston Center for Clinical Research, Sugar Land, Texas
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (12):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St. George Dermatology & Skin Care Centre, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - North Eastern Health Specialists, Hectorville, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Skin and Cancer Foundation, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Canada (16):
  - Institute for Skin Advancement, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - CCA Medical Research, Ajax, Ontario
  - Mediprobe Research, London, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research, Markham, Ontario
  - DermEdge, Mississauga, Ontario
  - York Dermatology Clinic and Research Centre, Mississauga, Ontario
  - Office of Dr. Niakosari Firouzeh, North York, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - Toronto Dermatology Centre, Toronto, Ontario
  - Dermatology on Bloor, Toronto, Ontario
  - Kim Papp Clinical Research, Waterloo, Ontario
  - Dr. Isabelle Delorme, Drummondville, Quebec
  - Innovaderm Research, Montreal, Quebec
- Czechia (8):
  - Nemocnice Jihlava, Jihlava
  - Nemocnice Novy Jicin a.s., Nový Jičín
  - MUDr. Helena Korandova, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Clintrial, Prague
  - Sanatorium profesora Arenbergera, Prague
  - Kozni a zilni ambulance, Ústí nad Labem
  - Krajska zdravotni - Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- Finland (3):
  - Terveystalo Tampere, Tampere
  - Mehilainen Turku, Turku
  - Local Institution - 0197, Vaasa
- France (4):
  - Hopital Prive dAntony, Antony
  - Centre Hospitalier Regional Universitaire Brest Hopital Morvan, Brest
  - Centre Hospitalier Universitaire de Nice Hopital lArchet, Nice
  - Centre Hospitalier Universitaire de Toulouse- Hopital Larrey, Toulouse
- Germany (13):
  - Local Institution - 0128, Augsburg
  - Hautarztpraxis Dr. Niesmann & Dr. Othlinghaus, Bochum
  - Hautarztpraxis Dr. Beatrice Gerlach, Dresden
  - Local Institution - 0246, Frankfurt am Main
  - Local Institution - 0119, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Dermakiel - Allergie Und Haut Centrum, Kiel
  - Praxis Dr. Beate Schwarz, Langenau
  - Universitatsklinikum Schleswig-Holstein - Campus Lubeck, Lübeck
  - Klinikum rechts der Isar der Technischen Universitat Munchen Klinik und Poliklinik fur Dermatolog, München
  - Harzklinikum Dorothea Christiane Erxleben, Quedlinburg
  - Praxis Dr. med. Wilfried Steinborn, Straubing
  - CentroDerm GmbH, Wuppertal
- Hungary (11):
  - Qualiclinic Egeszsegugyi Szolgaltato es Kutatasszervezo Kft., Budapest
  - Synexus Magyarorszag, Budapest
  - Semmelweis Egyetem, Budapest
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato - Debrecen Affiliated Site, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft. - Affiliated Site Gyula, Gyula
  - Josa Andras Oktatokorhaza - Szabolcs Szatmar-Bereg Megyei Onkormanyzat, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem, Szeged
  - Allergo-Derm Bakos, Szolnok
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato - Zalaegerszeg, Zalaegerszeg
- Israel (4):
  - Local Institution, Haifa
  - Local Institution, Kfar Saba
  - Local Institution, Petah Tikva
  - Local Institution, Ramat Gan
- Italy (2):
  - Azienda Ospedaliero Universitaria di Bologna Policlinico SantOrsola-Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Pisana Ospedale Santa Chiara, Pisa
- New Zealand (3):
  - Local Institution, Hamilton
  - Local Institution, Mount Cook
  - Local Institution, Tauranga
- Poland (17):
  - ZDROWIE OSTEO-MEDIC s.c. Lidia i Artur Racewicz, Agnieszka i Jerzy Supronik, Bialystok
  - ClinicMed Daniluk Nowak Spolka Jawna, Bialystok
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Synexus Polska Oddzial w Gdansk, Gda?sk
  - Zespol Naukowo-Leczniczy Iwolang, Iwonicz-Zdrój
  - Krakowskie Centrum Medyczne, Krakow
  - Dermed Centrum Medyczne, Lodz
  - Dermoklinika Centrum Medyczne S.C. M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej MED-LASER, Lublin
  - ETG - Siedlce, Siedlce
  - ETG - Skierniewice, Skierniewice
  - Local Institution - 0142, Torun
  - High-Med Przychodnia Specjalistyczna, Warsaw
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - ETG - Warszawa, Warsaw
  - Klinika Ambroziak, Warsaw
  - Local Institution - 0183, Wroclaw
- GCM Medical Group, San Juan, Puerto Rico
- Spain (9):
  - Local Institution - 0156, Córdoba
  - Hospital Universitario de Vinalopo, Elche
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital de Manises, Manises
  - Hospital Universitario Virgen de la Victoria, Mߧa
  - Local Institution - 0137, Pozuelo de Alarcón
  - Burbage Surgery, Santiago de Compostela
  - Consorci Hospital General Universitari de Valencia, Valencia
- Sweden (5):
  - Ladulaas Kliniska Studier, Borås
  - Pharmasite - Helsingborg, Helsingborg
  - ProbarE i Lund, Lund
  - PharmaSite - Malmo, Malmo
  - Karolinska Universitetssjukhuset, Solna
- United Kingdom (8):
  - MAC Clinical Research - Cannock, Cannock
  - Ashgate Medical Practice, Chesterfield
  - Local Institution - 0189, Chorley
  - Mounts Bay Medical, Cornwall
  - The Dudley Group NHS Foundation Trust, Dudley
  - MAC Clinical Research - Stockton, Durham
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - MAC Clinical Research - Manchester, Manchester

REFERENCES:
- [Derived] Armstrong AW, Warren RB, Sofen H, Spelman L, Linaberry M, Becker B, Jou YM, Daamen C, Kimball AB. Deucravacitinib in Plaque Psoriasis After Inadequate Response to Apremilast: Phase 3 POETYK Analysis. Dermatol Ther (Heidelb). 2025 Dec 5. doi: 10.1007/s13555-025-01606-9. Online ahead of print. PMID 41350512
- [Derived] Merola JF, Mease PJ, Armstrong AW, Strand V, Lehman T, Varga S, Choi JC, Becker B, Zhong Y, Colombo MJ, Thaci D, Bili A, Gottlieb AB. Deucravacitinib in Patients with Plaque Psoriasis Who Screened Positive for Psoriatic Arthritis: Improvements in Joint Pain and the Impact of Musculoskeletal Symptoms. Dermatol Ther (Heidelb). 2025 Aug;15(8):2281-2293. doi: 10.1007/s13555-025-01428-9. Epub 2025 May 30. PMID 40445270
- [Derived] Armstrong AW, Kircik L, Stein Gold L, Strober B, De Oliveira CHMC, Vaile J, Jou YM, Daamen C, Scharnitz T, Lebwohl M. Deucravacitinib: Laboratory Parameters Across Phase 3 Plaque Psoriasis Trials. Dermatol Ther (Heidelb). 2025 Apr;15(4):1025-1035. doi: 10.1007/s13555-025-01362-w. Epub 2025 Mar 20. PMID 40113724
- [Derived] Armstrong AW, Lebwohl M, Warren RB, Sofen H, Imafuku S, Ohtsuki M, Spelman L, Passeron T, Papp KA, Kisa RM, Vaile J, Berger V, Vritzali E, Hoyt K, Colombo MJ, Scotto J, Banerjee S, Strober B, Thaci D, Blauvelt A. Safety and Efficacy of Deucravacitinib in Moderate to Severe Plaque Psoriasis for Up to 3 Years: An Open-Label Extension of Randomized Clinical Trials. JAMA Dermatol. 2025 Jan 1;161(1):56-66. doi: 10.1001/jamadermatol.2024.4688. PMID 39602111
- [Derived] Armstrong AW, Augustin M, Beaumont JL, Pham TP, Hudgens S, Gordon KB, Zhuo J, Becker B, Zhong Y, Kisa RM, Banerjee S, Papp KA. Deucravacitinib Improves Patient-Reported Outcomes in Patients with Moderate to Severe Psoriasis: Results from the Phase 3 Randomized POETYK PSO-1 and PSO-2 Trials. Dermatol Ther (Heidelb). 2024 Aug;14(8):2235-2248. doi: 10.1007/s13555-024-01224-x. Epub 2024 Jul 30. PMID 39080153
- [Derived] Strober B, Thaci D, Sofen H, Kircik L, Gordon KB, Foley P, Rich P, Paul C, Bagel J, Colston E, Throup J, Kundu S, Sekaran C, Linaberry M, Banerjee S, Papp KA. Treatment of plaque psoriasis with deucravacitinib (POETYK PSO-2 study): a plain language summary. Immunotherapy. 2023 Aug;15(11):787-797. doi: 10.2217/imt-2023-0062. Epub 2023 May 7. PMID 37150956
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 Participant stopped treatment after week 16 and re-entered in treatment period Week 24-52.
Groups:
- BMS-986165: Participants receive 6 mg of BMS-986165 by oral administration once daily (QD).
  Participants originally randomized to BMS-986165 who are PASI 75 responders at Week 24 are re-randomized to BMS-986165 or placebo. Nonresponders at Week 24 will continue to receive BMS-986165 at Week 24.
- Placebo: Participants receive Placebo by oral administration once daily (QD).
  Participants originally randomized to placebo switch to BMS-986165 at Week 16.
- Apremilast: Participants receive 30 mg of Apremilast by oral administration twice daily (BID) (with initial titration per label)
  * 10 mg used for titration Day 1 through Day 3 morning dose
  * 20 mg used for titration Day 3 evening dose through Day 5 morning dose.
  * 30 mg from Day 5 evening dose onwards.
  Participants originally randomized to apremilast who are PASI 75 responders at Week 24 are switched to placebo at Week 24. Nonresponders at Week 24 are switched to BMS-986165 at Week 24.
Period: Pre-treatment
Arm/Group | BMS-986165 | Placebo | Apremilast
Started | 511 | 255 | 254
Completed | 510 | 254 | 254
Not Completed | 1 | 1 | 0
Not completed — Randomized but not treated | 1 | 1 | 0
Period: Treatment Week 0 - Week 16
Arm/Group | BMS-986165 | Placebo | Apremilast
Started | 510 | 254 | 254
Completed | 456 | 212 | 217
Not Completed | 54 | 42 | 37
Not completed — Adverse Event | 11 | 7 | 12
Not completed — Lack of Efficacy | 6 | 9 | 4
Not completed — Lost to Follow-up | 5 | 6 | 2
Not completed — Non-compliance with protocol | 5 | 2 | 1
Not completed — Withdrawal by Subject | 14 | 9 | 9
Not completed — Other reasons | 13 | 9 | 7
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Period: Treatment Week 16 - Week 24
Arm/Group | BMS-986165 | Placebo | Apremilast
Started | 667 | 0 | 217
Completed | 642 | 0 | 208
Not Completed | 25 | 0 | 9
Not completed — Adverse Event | 7 | 0 | 2
Not completed — Lack of Efficacy | 8 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Non-compliance with protocol | 3 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Other reasons | 2 | 0 | 3
Not completed — Pregnancy | 1 | 0 | 1
Period: Treatment Week 24 - Week 52
Arm/Group | BMS-986165 | Placebo | Apremilast
Started | 604 | 247 | 0
Completed | 535 | 214 | 0
Not Completed | 69 | 33 | 0
Not completed — Adverse Event | 14 | 7 | 0
Not completed — Lack of Efficacy | 8 | 8 | 0
Not completed — Lost to Follow-up | 9 | 4 | 0
Not completed — Non-compliance with protocol | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 0
Not completed — Other reasons | 28 | 7 | 0
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986165 | Placebo | Apremilast | Total
Number analyzed (Participants) | 511 | 255 | 254 | 1020
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (13.37) | 47.3 (13.57) | 46.4 (13.28) | 46.9 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 74 | 97 | 346
  Male | 336 | 181 | 157 | 674
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 29 | 29 | 116
  Not Hispanic or Latino | 445 | 226 | 223 | 894
  Unknown or Not Reported | 8 | 0 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 474 | 232 | 229 | 935
  Black or African American | 8 | 9 | 9 | 26
  Asian | 24 | 8 | 12 | 44
  American Indian or Alaska Native | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 3 | 4 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Static Physician's Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (sPGA 0/1)
Description: The sPGA is a 5-point scale average assessment of all psoriatic lesions graded for erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as: clear (0), almost clear (1), mild (2), moderate (3), or severe (4). The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. The higher sPGA score denotes to more severe disease activity. sPGA 0/1 is the response as a number of participants who experience a sPGA score that determines psoriasis severity as 0 or 1 with at least a 2-point improvement from baseline using the non-responder imputation (NRI) method.
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants in the BMS-986165 and Placebo arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 511 | 255
Participants | 253 | 22
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 10.55, 95% CI 2-sided [6.54 to 17.00]

2. Primary Outcome: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (PASI 75)
Description: The Psoriasis Area and Severity Index (PASI) is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance.
  The PASI is a measure of the average erythema (redness), infiltration (thickness), and desquamation (scaling) of psoriatic skin lesions (each graded on a 0-4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the response as a number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method. Baseline is defined as the measurement at the randomization visit (Week 0).
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Baseline and Week 16
Population: All randomized participants in the BMS-986165 and Placebo arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 511 | 255
Participants | 271 | 24
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 10.49, 95% CI 2-sided [6.65 to 16.55]

3. Secondary Outcome: The Number of Participants Who Achieve a 90% Improvement From Baseline in the Psoriasis Area and Severity Index Score at Week 16 (PASI 90)
Description: The Psoriasis Area and Severity Index (PASI) is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance.
  The PASI is a measure of the average erythema (redness), infiltration (thickness), and desquamation (scaling) of psoriatic skin lesions (each graded on a 0-4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 is the response as a number of participants who experience at least a 90% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method. Baseline is defined as the measurement at the randomization visit (Week 0).
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Baseline and Week 16
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 511 | 255 | 254
Participants | 138 | 7 | 46
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 11.42, 95% CI 2-sided [5.45 to 23.93]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.18 to 2.56]

4. Secondary Outcome: The Number of Participants Who Achieve a 100% Improvement From Baseline in the Psoriasis Area and Severity Index Score at Week 16 (PASI 100)
Description: The Psoriasis Area and Severity Index (PASI) is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance.
  The PASI is a measure of the average erythema (redness), infiltration (thickness), and desquamation (scaling) of psoriatic skin lesions (each graded on a 0-4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 100 is the response as a number of participants who experience at least a 100% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method. Baseline is defined as the measurement at the randomization visit (Week 0).
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Baseline and Week 16
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 511 | 255 | 254
Participants | 52 | 3 | 11
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 9.21, 95% CI 2-sided [2.89 to 29.40]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0051, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.30 to 5.00]

5. Secondary Outcome: The Number of Participants With a Static Physician Global Assessment Score of 0 at Week 16 (sPGA 0)
Description: The sPGA is a 5-point scale average assessment of all psoriatic lesions graded for erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as: clear (0), almost clear (1), mild (2), moderate (3), or severe (4). The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. sPGA 0 is the response as a number of participants who experience a sPGA score that determines psoriasis severity as 0 using the non-responder imputation (NRI) method.
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 511 | 255 | 254
Participants | 80 | 3 | 16
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 14.44, 95% CI 2-sided [4.62 to 45.11]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.85, 95% CI 2-sided [1.61 to 5.03]

6. Secondary Outcome: Change From Baseline in Psoriasis Symptoms and Signs Diary (PSSD) Symptom Score at Week 16
Description: PSSD assesses the severity of 5 symptoms (itch, pain, stinging, burning, skin tightness) and 6 participant-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding). The severity of each item is rated on an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). Both symptom and sign scores are derived by averaging the questions and multiplying by 10. A total PSSD score ranging 0-100 will be derived from taking the average of the symptom and sign scores. 0 represents the least severe symptom/sign and 100 represents the most severe. Baseline is defined as the measurement at the randomization visit (Week 0).
  A modified observation carried forward (mBOCF) approach will be used for missing data. The baseline observation will be carried forward for participants who discontinue study treatment for all analysis weeks after the assessment time point of discontinuation due to lack of efficacy and AEs.
Time Frame: Baseline and Week 16
Population: All randomized participants with evaluable baseline and week 16 PSSD scores.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 466 | 239 | 233
Score on a scale | -28.9 (25.22) | -4.2 (19.58) | -21.5 (25.44)
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = -23.6, 95% CI 2-sided [-26.9 to -20.3], Standard Error of Mean 1.67
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = -7.2, 95% CI 2-sided [-10.5 to -3.9], Standard Error of Mean 1.68

7. Secondary Outcome: Psoriasis Symptoms and Signs Diary (PSSD) Symptom Score of 0 at Week 16
Description: Psoriasis Symptoms and Signs Diary (PSSD) is an 11-item participant-reported instrument that assesses severity of symptoms and participant-observed signs commonly associated in plaque psoriasis. The PSSD assesses severity of 5 symptoms (itch, pain, stinging, burning, skin tightness) and 6 participant-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding) using 0 to 10 numerical ratings. The severity of each item is rated on an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable) where the symptoms summary score is derived from the average of the scores. A higher score indicates more severe disease. PSSD 0 is the response as a number of participants who experience a PSSD symptom score that determines psoriasis severity as 0 among participants with a baseline PSSD symptom score >= 1 using the non-responder imputation (NRI) method.
Time Frame: Week 16
Population: All randomized participants with a baseline PSSD symptom score ≥ 1
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 466 | 238 | 232
Participants | 35 | 3 | 10
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.40, 95% CI 2-sided [1.94 to 21.15]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0928, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.89 to 3.71]

8. Secondary Outcome: The Number of Participants With a Scalp Specific Physician's Global Assessment (Ss-PGA) Score 0 or 1 at Week 16 (Ss-PGA 0/1)
Description: The scalp specific Physician's Global Assessment (ss-PGA) evaluates scalp lesions in terms of clinical signs of redness, thickness, and scaliness and scored on the following 5-point ss-PGA scale: 0 = absence of disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, 4 = severe disease. ss-PGA 0/1 is the response as a number of participants who experience a ss-PGA score of 0 or 1 with at least a 2-point improvement from baseline among participants with a baseline ss-PGA score ≥3 .
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants with a baseline ss-PGA score >=3
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 305 | 173 | 166
Participants | 182 | 30 | 61
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.85, 95% CI 2-sided [4.34 to 10.81]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.77 to 3.91]

9. Secondary Outcome: The Number of Participants With a Dermatology Life Quality Index (DLQI) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (DLQI 0/1)
Description: The DLQI is a participant-reported quality of life index which consists of 10 questions concerning how much skin problems affect symptoms and feelings, daily activities, leisure, work, school, personal relationships, and treatment during the last week. Each question is scored on a scale of 0 to 3 where 0 = not at all, 1 =a little, 2 = a lot, or 3 = very much. The scores are summed, giving a range from 0 (no impairment of life quality) to 30 (maximum impairment). DLQI 0/1 is the number of participants with a score of 0 or 1 among participants with a baseline DLQI score ≥2.
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants with a baseline DLQI score >=2. Pre-specified for data to be collected only in BMS-986165 and Placebo arms.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 495 | 246
Participants | 186 | 24
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.38, 95% CI 2-sided [3.42 to 8.47]

10. Secondary Outcome: The Number of Participants With a Physician Global Assessment- Fingernails (PGA-F) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (PGA-F 0/1)
Description: The Physician Global Assessment- Fingernails (PGA-F) evaluates the overall condition of the fingernails and is rated on a 5-point scale:0 = clear, 1 = minimal, 2 = mild, 3 = moderate, and 4 = severe. PGA-F 0/1 is the response as a number of participants with a PGA-F score of 0 or 1 with at least a 2-point improvement from baseline among participants with a baseline PGA-F score >=3.
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants with a baseline PGA-F score >=3. Pre-specified for data to be collected only in BMS-986165 and Placebo arms.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 69 | 38
Participants | 14 | 3
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p = 0.0621, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.21, 95% CI 2-sided [0.88 to 11.79]

11. Secondary Outcome: The Number of Participants With a Palmoplantar Physician's Global Assessment (Pp-PGA) Score of 0 or 1 at Week 16 (Pp-PGA 0/1)
Description: The palmoplantar Physician's Global Assessment (pp-PGA) score evaluates palmoplantar (including finger and toe surfaces) psoriasis lesions based on overall severity by investigator, then scored on the following 5-point scale: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; and 4 = severe. pp-PGA 0/1 is the number of participants with a score of 0 or 1 among participants with a baseline pp-PGA score ≥ 3.
Time Frame: Week 16
Population: All randomized participants with a baseline pp-PGA score >=3.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 39 | 17 | 20
Participants | 18 | 4 | 8
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p = 0.6692, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.06 to 7.46]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.3793, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.02 to 5.56]

12. Secondary Outcome: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 16 (PASI 75)
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: All randomized participants in the BMS-986165 and Apremilast arms.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 511 | 254
Participants | 271 | 101
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.29 to 2.41]

13. Secondary Outcome: The Number of Participants With a Static Physician Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Apremilast at Week 16 (sPGA 0/1)
Description: The sPGA is a 5-point scale average assessment of all psoriatic lesions graded for erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as: clear (0), almost clear (1), mild (2), moderate (3), or severe (4). The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. sPGA 0/1 is the number of participants with a sPGA score of 0 or 1 with at least a 2-point improvement from baseline.
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 16 or who have missing Week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants in the BMS-986165 and Apremilast arms.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 511 | 254
Participants | 253 | 86
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.45 to 2.78]

14. Secondary Outcome: Time to Relapse Until Week 52 Among Week 24 PASI 75 Responders
Description: Relapse is defined as 50% loss or greater of Week 24 PASI percent improvement from baseline.
  The PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0-4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity.
Time Frame: From Week 24 to Week 52 (up to approximately 28 weeks)
Population: All randomized participants who had PASI 75 response at week 24. Pre-specified to report participants from their original randomization.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 145 | 150 | 95
Days | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 197.0 [125.0 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Log Rank

15. Secondary Outcome: The Number of Participants With a Static Physician Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Apremalist at Week 24 (sPGA 0/1)
Description: The sPGA is a 5-point scale average assessment of all psoriatic lesions graded for erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as: clear (0), almost clear (1), mild (2), moderate (3), or severe (4). The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. sPGA 0/1 is the number of participants with a sPGA score of 0 or 1.
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 24 or who have missing Week 24 endpoint data for any reason.
Time Frame: Week 24
Population: All randomized participants. Pre-specified for data to be collected only in the BMS-986165 and Apremilast arms and from participants original randomization. Participants who had any visit impacted by COVID will be excluded from that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 504 | 254
Participants | 251 | 75
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.78 to 3.43]

16. Secondary Outcome: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Apremalist at Week 24 (PASI 75)
Description: The Psoriasis Area and Severity Index (PASI) is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance.
  PASI is a measure of the average erythema (redness), infiltration (thickness), and desquamation (scaling) of psoriatic skin lesions (each graded on a 0-4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the response as a number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method. Baseline is defined as the measurement at the randomization visit (Week 0).
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 24 or who have missing Week 24 endpoint data for any reason.
Time Frame: Baseline and Week 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 504 | 254
Participants | 296 | 96
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.78 to 3.36]

17. Secondary Outcome: The Number of Participants Who Achieve a 90% Improvement From Baseline in the Psoriasis Area and Severity Index Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 24 (PASI 90)
Description: The Psoriasis Area and Severity Index (PASI) is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance.
  PASI is a measure of the average erythema (redness), infiltration (thickness), and desquamation (scaling) of psoriatic skin lesions (each graded on a 0-4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 is the response as a number of participants who experience at least a 90% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method. Baseline is defined as the measurement at the randomization visit (Week 0).
  Non-responder imputation (NRI) will be used for participants who: Discontinue treatment or study prior to Week 24 or who have missing Week 24 endpoint data for any reason.
Time Frame: Baseline and week 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 504 | 254
Participants | 164 | 50
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.43 to 3.01]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from their first dose until the study was completed (up to approximately 60 weeks). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 56 weeks)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- BMS-986165 (Week 0 up to Week 16); BMS-986165 (Week 0 up to Week 52): Participants receive 6 mg of BMS-986165 by oral administration once daily (QD)
- Placebo (Week 0 up to Week 16); Placebo (Week 0 up to Week 52): Participants receive Placebo by oral administration once daily (QD)
- Apremilast (Week 0 up to Week 16); Apremilast (Week 0 up to Week 52): Participants receive 30 mg of Apremilast by oral administration twice daily (BID) (with initial titration per label)
  10 mg used for titration Day 1 through Day 3 morning dose
  20 mg used for titration Day 3 evening dose through Day 5 morning dose.
  30 mg from Day 5 evening dose onwards
Arm/Group | BMS-986165 (Week 0 up to Week 16) | Placebo (Week 0 up to Week 16) | Apremilast (Week 0 up to Week 16) | BMS-986165 (Week 0 up to Week 52) | Placebo (Week 0 up to Week 52) | Apremilast (Week 0 up to Week 52)
All-Cause Mortality (participants affected / at risk) | 1/511 | 0/255 | 1/254 | 2/834 | 0/502 | 1/254
Serious Adverse Events (participants affected / at risk) | 8/510 | 3/254 | 1/254 | 24/833 | 5/501 | 3/254
Other Adverse Events (participants affected / at risk) | 114/510 | 61/254 | 86/254 | 249/833 | 97/501 | 98/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 (Week 0 up to Week 16) (N=510) | Placebo (Week 0 up to Week 16) (N=254) | Apremilast (Week 0 up to Week 16) (N=254) | BMS-986165 (Week 0 up to Week 52) (N=833) | Placebo (Week 0 up to Week 52) (N=501) | Apremilast (Week 0 up to Week 52) (N=254)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Mycoplasma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0
Purulence (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Vascular graft infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malignant hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 (Week 0 up to Week 16) (N=510) | Placebo (Week 0 up to Week 16) (N=254) | Apremilast (Week 0 up to Week 16) (N=254) | BMS-986165 (Week 0 up to Week 52) (N=833) | Placebo (Week 0 up to Week 52) (N=501) | Apremilast (Week 0 up to Week 52) (N=254)
Diarrhoea (Gastrointestinal disorders) | 24 | 19 | 33 | 39 | 22 | 35
Nausea (Gastrointestinal disorders) | 7 | 3 | 23 | 13 | 6 | 26
Nasopharyngitis (Infections and infestations) | 55 | 29 | 23 | 133 | 47 | 28
Upper respiratory tract infection (Infections and infestations) | 25 | 11 | 14 | 74 | 27 | 21
Headache (Nervous system disorders) | 22 | 14 | 28 | 45 | 16 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03611751/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03611751/SAP_001.pdf